CLINICAL TRIAL: NCT04785846
Title: Prospective, Single-arm, Multicenter, Observational, Prospective Registry of RESOLUTE-ONYX™ Zotarolimus-eluting Stent Utilization in Percutaneous Small Vessel Coronary Interventionism.
Brief Title: Registry of RESOLUTE-ONYX™ Zotarolimus-eluting Stent Utilization in Percutaneous Small Vessel Coronary Interventionism.
Acronym: Disco-9
Status: Completed | Type: Observational
Sponsor: Fundación Investigación Sanitaria en León (Other)
Responsible Party: Sponsor
Other Study IDs: Disco 9
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Coronary Disease; Angina, Stable; Ischemia; Acute Coronary Syndrome; Percutaneous Coronary Intervention
Keywords: Small vessels; Coronary Disease; Angina, Stable; Ischemia; Acute Coronary Syndrome; Percutaneous Coronary Intervention; Stent
MeSH Terms: conditions — Coronary Disease; Angina, Stable; Ischemia; Acute Coronary Syndrome | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Single Group: Adult patients with coronary artery disease undergoing percutaneous coronary intervention on vessels with a diameter less than or equal to 2.5 mm.
  Interventions: Device: Percutaneous Coronary Intervention

INTERVENTIONS:
Device: Percutaneous Coronary Intervention — Percutaneous Coronary Intervention

SUMMARY:
DESIGN: Prospective, single-arm, multicenter, observational, prospective registry of the use of the RESOLUTE-ONYX™ zotarolimus-eluting stent in percutaneous coronary intervention in small vessels.

Clinical follow-up at 1 month, 6 months and 1 year.

OBJECTIVE: To evaluate the safety and efficacy of using RESOLUTE-ONYX zotarolimus-eluting stent in PCI in small vessels (diameter ≤2.5 mm).

DISEASE UNDER STUDY: Adult patients with coronary artery disease (stable angina, silent ischemia or non-ST-segment elevation acute coronary syndrome) undergoing percutaneous coronary intervention on vessels with a diameter less than or equal to 2.5 mm.

TOTAL NUMBER OF PATIENTS: Approximately 320 patients are expected to be included in the study.

DETAILED DESCRIPTION:
1.1 STUDY TITLE:

Prospective, single-arm, multicenter, observational, prospective registry of use of the RESOLUTE-ONYX™ zotarolimus-eluting stent in percutaneous small vessel coronary intervention (DISCO 9 study).

1.2 SPONSOR:

Fundación de Investigación Sanitaria en León (FISLeón) Complejo Asistencial Universitario de León.

Altos de Nava s/n 24008 León. SPAIN.

1.3 COORDINATING RESEARCHER OF THE STUDY

Dr. Juan Carlos Cuellas Ramón Section of Hemodynamics and Interventional Cardiology. Cardiology Service. Cardiology Service.

Complejo Asistencial Universitario de León.

1.4 OBJECTIVE:

To evaluate the safety and efficacy of using RESOLUTE-ONYX zotarolimus-eluting stent in PCI in small vessels (diameter ≤2.5 mm).

1.5 PRIMARY ENDPOINT:

Incidence of Major Adverse Cardiac Events (MACE) defined as a composite of: death of cardiac origin, target vessel-related myocardial infarction and/or new target lesion revascularization (percutaneous or surgical) assessed at 1 year.

1.6 SECONDARY ENDPOINTS:

* Procedure success.
* Periprocedural myocardial infarction.
* Each of the separate components of the combined event: death of cardiac origin, target vessel-related myocardial infarction, new target lesion revascularization (percutaneous or surgical) assessed at 1 month, 6 months, 1 year.
* Acute/sub-acute thrombosis (definite/probable according to ARC definitions, Appendix 2).
* Bleeding unrelated to surgical revascularization. Classification of BARC bleeding .
* Duration of dual antiplatelet therapy.

1.7 INCLUSION CRITERIA

* Signed written Informed Consent.
* Patients over 18 years of age.
* Males or post-menopausal women or women under contraceptive treatment. Women of childbearing age must have a negative pregnancy test.
* Diagnosis of stable angina, silent ischemia or non-ST-segment elevation acute coronary syndrome (unstable angina or non-Q infarction).
* De novo coronary artery disease, single-vessel or multivessel, with stenosis >70% according to visual estimation, susceptible to treatment with intracoronary stenting.
* Coronary stenosis affects a vessel with diameter ≥2 mm and ≤2.5 mm.
* The implantation of the RESOLUTE-ONYX™ zotarolimus-eluting stent used according to the indications for use in routine clinical practice at the center.

1.8 EXCLUSION CRITERIA

* Acute myocardial infarction with ST-segment elevation during the hospitalization in which the patient is included.
* Significant left main coronary artery stenosis.
* In-stent restenosis.
* Chronic total occlusion.
* Stenosis in aorto-coronary grafts of saphenous vein or mammary or radial artery.
* Hemorrhagic diathesis or high risk of bleeding.
* Treatment with oral anticoagulants.
* Allergy to aspirin, clopidogrel, prasugrel or ticagrelor.
* Known allergy to zotarolimus, nickel, chromium or cobalt.
* Women who are pregnant, breastfeeding or expect to become pregnant within the next year.
* Participation in another clinical study.
* Limited life expectancy (< 1 year).
* Planned major elective surgery.
* Inability to complete follow-up.

1.9 DISEASE UNDER STUDY

Adult patients with coronary artery disease (stable angina, silent ischemia or non-ST-segment elevation acute coronary syndrome) undergoing percutaneous coronary intervention on vessels with a diameter less than or equal to 2.5 mm.

1.10 DEVICE

Medical device with CE marking and approved indication and commonly used in participating hospitals.

1.11 TOTAL NUMBER OF PATIENTS

Approximately 320 patients are expected to be included in the study.

1.12 SELECTION METHOD

Patients with coronary artery disease and stable angina, silent ischemia or non-ST-segment elevation acute coronary syndrome (unstable angina or non-Q infarction) who are going to undergo PCI and who have stenoses to be treated in vessels with a diameter equal to or less than 2.5mm.

1.13 METHOD OF EVALUATION

Major adverse cardiac events will be analyzed, which are defined as:

* Death of cardiac origin.
* Nonfatal infarction related to the target vessel. Definitions according to the third universal definition of myocardial infarction.
* New revascularization of the target lesion.

In addition, the following will be analyzed:

* Stent thrombosis. Definitions according to the ARC (Academic Research Consortium).
* Bleeding not related to surgical revascularization. Classification of BARC bleeding

1.14 REGISTRATION SYSTEM

The data collection notebook (eCRD) will be in electronic format. The database with on-line collection will be prepared by the company in charge of managing the study (CRO). Each variable to be collected will have a field where the information will be entered manually or one of the options available for the field in question will be chosen.

1.15 PROCEDURE

The procedure will be performed according to each site's standard practice. The lesion will be treated with a RESOLUTE- ONYX™ zotarolimus-eluting stent of 2, 2.25 or 2.5 mm in diameter. The choice, by the operator, of stent size and length will be made according to visual estimation. The need for additional stents will be at the operator's discretion but they should always be RESOLUTE-ONYX™ in the same lesion. Direct stenting is recommended. The need for predilatation or postdilatation and the balloons used will be at the operator's discretion.

An attempt should be made to achieve a stent to artery diameter ratio of 1.1 to 1.2 to 1.1. 1.2 to 1. The procedure will be considered successful when the device is implanted with a residual stenosis of less than 20% and TIMI 3 flow in the treated vessel.

In cases of multivessel disease, RESOLUTE-ONYX™ stents will always be used in lesions in vessels with diameters less than or equal to 2.5 mm, even if performed at different times. In the case of stenosis in vessels of 2.75 mm or more, the stents considered appropriate by the operator will be used, although it is recommended that if a DES is chosen, it should be zotarolimus-eluting.

The access route can be radial or femoral. Antiplatelet therapy and anticoagulation will be performed according to the clinical practice guidelines (http://www.escardio.org/GUIDELINES-SURVEYS/Pages/welcome.aspx) and the protocols established in each center. It is recommended to take into account the bleeding risk according to the CRUSADE scale score. Double antiplatelet therapy and its maintenance time will be performed according to the clinical practice guidelines and protocols of the center. Doses of unfractionated heparin or low molecular weight heparin during the procedure and the use of bivalirudin or abciximab will be at the operator's discretion. The drugs used and their dosage will be recorded.

Medical treatment at discharge will be at the discretion of the corresponding cardiologist following clinical practice guidelines. In diabetic or prediabetic patients, fasting blood glucose (>8h) and glycated hemoglobin A1C will be determined during admission, according to hospital practice, for the management of these patients as described in the clinical practice guidelines.

Clinical follow-up, once discharged, will be carried out by telephone or in person at 30 days, 6 months and 12 months.

1.16 STATISTICAL ANALYSIS

Statistical analysis will be performed with SPSS software in the most current version available at the time of analysis.

Sample size calculation

If we estimate that the proportion of MACE per year with zotarolimus stents in small vessel PCI is 8-10% and the best published observed outcome, in this case with everolimus stents, is 4%, data expected to be achieved with the stent used in this observational registry, assuming a risk of 5% and a ß 20% risk with a bilateral contrast and a 10% loss to follow-up, we would need to include 320 patients to demonstrate this difference.

Data processing

A study-specific data management plan will be prepared defining all aspects of data management and processing. This data management plan will include in detail:

* Validation processes.
* Query resolution process.
* Structure and fundamental parts of the study data collection application.
* General data considerations including validation rules and normality ranges used for the different parameters collected in the study.

The data will be stored in a relational database on a MySQL server. The application will be duly protected by means of a SSL security certificate for the correct encryption of the transferred data.

Data analysis

Discrete variables will be described by providing frequency and percentage. For the description of continuous variables, the mean, median, standard deviation, minimum and maximum will be used. The incidence of MACE at 1 month, 6 months and 1 year, will be described by frequency and percentage in each of the periods indicated.

Differences between proportions will be analyzed according to test 2. Differences between discrete and continuous variables according to t-Student or ANOVA (for discrete variables of several categories) and the comparison between two continuous variables with a regression model, if the distributions are normal, or the respective nonparametric tests, if they are not.

Event-free survival is defined as the time elapsed from the time the patient enters the study until the first major cardiovascular event occurs. A Kaplan Meyer analysis will be performed for event-free survival presenting the number of events, censored and median event-free survival and its 95% confidence interval.

A logistic regression analysis will be performed to determine those possible factors that may determine the occurrence of a cardiovascular event at 12 months. For the construction of the model, those variables considered potentially influential under clinical criteria will be selected.

1.17 ADVERSE EVENTS

For the purposes of this protocol, an adverse event is any undesirable medical episode that occurs in a patient. This definition is not dependent on causal relationship to the stent or protocol requirements.

If it is established that an adverse event has occurred, the investigator should obtain all the information necessary to complete the adverse event form in the data collection form.

Given the characteristics of this study, only those AA that, in the opinion of the investigator, are relevant and/or related to the therapy under study will be collected

1.18 SERIOUS ADVERSE EVENTS (SAEs)

All serious adverse events should be reported to the sponsor within 24 hours of the investigator becoming aware of the event.

An adverse event is considered serious if:

* Causes death
* Produces a serious deterioration in the patient's health, which:

  * Causes a life-threatening injury or illness.
  * Causes permanent impairment of a bodily structure or function
  * Requires hospitalization of the patient or a prolongation of hospitalization, if already hospitalized
  * Requires medical or surgical intervention to prevent permanent impairment of a body structure or function permanent impairment of a bodily structure or function
  * In addition, any major adverse cardiac event (MACE) Requires notification within 24 hours.

All serious adverse events should be followed up until they are resolved (with or without sequelae).

1.19 INFORMED CONSENT

Before being admitted to the study and in accordance with current regulations, the patient must give written consent to participate in the study, once he/she has been informed of the nature, scope and possible consequences of the study in a language understandable to him/her.

1.20 GENERAL CONSIDERATIONS

In this study, the standards of good clinical practice (GCP) applicable to epidemiological studies will be followed to ensure that the design, conduct and communication of the data are reliable and that the rights and integrity of the participating subjects are protected while maintaining the confidentiality of their data, in accordance with EU directives, the Declaration of Helsinki and local regulations.

1.21 ETHICAL COMMITTEES

The study protocol will be submitted to the Clinical Research Ethics Committee (C.E.I.C.) of the Complejo Asistencial Universitario de León (CAULE) (National Coordinating Center of the study) for approval before initiating the study.

The modifications of the protocol as well as those of the patient information sheet and informed consent will be sent to the CEIC to obtain its approval before its application.

ELIGIBILITY:
Inclusion Criteria:

1. Signature of the Informed Consent in writing.
2. Patients over 18 years of age.
3. Males or post-menopausal women or women under contraceptive treatment. Women of childbearing age must have a negative pregnancy test.
4. Diagnosis of stable angina, silent ischemia or non-ST-segment elevation acute coronary syndrome (unstable angina or non-Q infarction).
5. De novo coronary artery disease, single-vessel or multivessel, with stenosis >70% according to visual estimation, susceptible to treatment with intracoronary stenting.
6. Coronary stenosis involving a vessel with diameter ≥2 mm and ≤2.5 mm.
7. Implantation of the RESOLUTE-ONYX™ zotarolimus-eluting stent used according to the indications for use in routine clinical practice at the center.

Exclusion Criteria:

1. Acute myocardial infarction with ST-segment elevation during the hospitalization in which the patient is included.
2. Significant stenosis of the left coronary artery trunk.
3. In-stent restenosis.
4. Chronic total occlusion.
5. Stenosis in aorto-coronary grafts of saphenous vein or mammary or radial artery.
6. Hemorrhagic diathesis or high risk of bleeding.
7. Treatment with oral anticoagulants.
8. Allergy to aspirin, clopidogrel, prasugrel or ticagrelor.
9. Known allergy to zotarolimus, nickel, chromium, or cobalt.
10. Women who are pregnant, breastfeeding or expect to become pregnant within the next year.
11. Participation in another clinical study.
12. Limited life expectancy (< 1 year).
13. Planned major elective surgery
14. Unable to complete follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with coronary artery disease (stable angina, silent ischemia or non-ST-segment elevation acute coronary syndrome) undergoing percutaneous coronary intervention on vessels with a diameter less than or equal to 2.5 mm.
Sampling Method: Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardiac Events (MACE) | 1 year
  Incidence of Major Adverse Cardiac Events (MACE) defined as a composite of: death of cardiac origin, target vessel-related myocardial infarction and/or new target lesion revascularization (percutaneous or surgical).

SECONDARY OUTCOMES:
Success of the procedure | In the procedure
  Success of the procedure
Periprocedural myocardial infarction | In the procedure
  Periprocedural myocardial infarction
Each of the separate components of the combined event: Death of cardiac origin, target vessel-related myocardial infarction, new target lesion revascularization (percutaneous or surgical) | 1 month, 6 months, 1 year.
  Each of the separate components of the combined event: Death of cardiac origin, target vessel-related myocardial infarction, new target lesion revascularization (percutaneous or surgical)
Acute/sub-acute thrombosis | 1 month, 6 months, 1 year
  Acute/sub-acute thrombosis (definite/probable according to ARC definitions)
Bleeding unrelated to surgical revascularization | 1 month, 6 months, 1 year
  Bleeding unrelated to surgical revascularization. Classification of BARC bleeding
Duration of dual antiplatelet therapy | 1 month, 6 months, 1 year
  Duration of dual antiplatelet therapy

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Cuellas Ramón, MD, Study Director — Fundación de Investigación Sanitaria de León
Locations (15):
- Spain (15):
  - University Hospital of Santiago de Compostela, Santiago de Compostela, A Coruña
  - University Hospital of Cruces, Barakaldo, Bizkaia
  - University Hospital Marqués de Valdecilla, Santander, Cantabria
  - University Hospital San Pedro, Logroño, La Rioja
  - University Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - University Hospital of Cabueñes, Gijón, Principality of Asturias
  - University Hospital of Canarias, San Cristóbal de La Laguna, Tenerife
  - University Hospital of Torrecárdenas, Almería
  - University Hospital Infanta Cristina, Badajoz
  - University Hospital Juan Ramón Jiménez, Huelva
  - León University Health Care Complex, León
  - University Hospital Virgen de la Victoria, Málaga
  - University Hospital Virgen de la Arrixaca, Murcia
  - University Hospital Miguel Servet, Zaragoza
  - University Hospital Txagorritxu, Vitoria-Gasteiz, Álava

IPD SHARING:
Plan to Share IPD: No